CLINICAL TRIAL: NCT06679179
Title: Effect of Flozin (dapagliflozin) Administration on Myocardial and Peripheral Vascular Remodeling
Acronym: DAPA-REMO
Status: Recruiting | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arkadiusz Niklas, Poznan University of Medical Sciences, Poznan University of Medical Sciences
Other Study IDs: 199/23
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to assess the effect of treatment with flozin (dapagliflozin 10mg once a day) on haemodynamic parameters and myocardial and peripheral vascular remodeling in patients with NYHA class II-III heart failure.

DETAILED DESCRIPTION:
In the available literature, there are reports of beneficial effects of flozins on improving myocardial systolic and diastolic function and isolated reports of effects on regression of organ damage (heart, vessels). These drugs significantly improve the prognosis of patients with heart failure, reduce total and cardiovascular mortality, reduce the number of exacerbations and the need for hospitalization, and have a beneficial effect on improving quality of life regardless of coexisting diabetes. New properties demonstrating the pleiotropic effect of the flozins are constantly being discovered. Drugs in this group are highly potent, selective and reversible inhibitors of the sodium ion-dependent glucose cotransporter 2 (SGLT2). The flozins have a low risk of side effects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed heart failure NYHA class II and III
* consent to participate in the study
* patients should already be receiving treatment with an ACE inhibitor or sacubitril/valsartan or sartans, a beta-blocker, and an MRA, and should start on SGLT2i as part of therapy enhancement

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over 18 years of age of both sexes with diagnosed heart failure NYHA class II and III.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Identify factors that predict remodeling and enhancement of left ventricular (LV) systolic and diastolic function within 12 months. | 6 months
  This study aims to identify factors that predict the remodeling and enhancement of left ventricular (LV) systolic and diastolic functions over 12 months. Using both univariate and multivariate logistic regression analyses, it will focus on finding predictors at the 6-month mark, especially through advanced echocardiography parameters and vascular stiffness test.

SECONDARY OUTCOMES:
Assessment of the combined outcome including deaths from cardiovascular causes, defibrillator discharges, hospitalizations or episodes of atrial fibrillation. | Baseline ut to 12 months
  Over 12 months, the study will assess a combined outcome including cardiovascular-related deaths, defibrillator discharges, hospitalizations, or atrial fibrillation episodes. Predictors for these cardiovascular events will be analyzed using univariate and multivariate Cox analyses, with the model's quality evaluated by time-dependent ROC analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Niklas, PhD, Principal Investigator — University Clinical Hospital in Poznań, 49 Przybyszewskiego Street, 60-355 Poznań
Locations (1):
- University Clinical Hospital in Poznań, 49 Przybyszewskiego Street, 60-355 Poznań, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No